Cover letter:

Official project title:

Efficacy of Mediterranean-DASH Intervention for Neurodegenerative Delay (MIND) Plus Forest Bathing (FB) on blood pressure and cognitive health for those who are aged 50 and above with hypertension

Funding source: N&HS Mini Grant

Project ethical approval number: HE-NHS2021/02

Document updated date: 20/04/2022

Document updated date: 20/04/2022

## **Information Sheet**

#### TITLE OF THE STUDY

Effect of Mediterranean-DASH Intervention for Neurodegenerative Delay (MIND) Plus Forest Bathing (FB) on blood pressure and cognitive health for those who are aged 50 and above with hypertension.

#### INTRODUCTORY SENTENCE

You are invited to participate in a research study conducted by Associate Professor, Dr. Law Pui Sze Queenie from the School of Nursing and Health Studies of the Hong Kong Metropolitan University (HKMU).

## PURPOSE OF THE STUDY

This study will aim to investigate the effect of MIND, MIND plus FB and usual-care control on hypertension. The result may provide indication to health care professionals and population at risk to integrate MIND or/and FB into the management of hypertension.

#### **PROCEDURES**

The study would be last for twelve weeks. You are invited to screen for the inclusion criteria and sign a consent form before participation in this study. You are invited to measure systolic BP, finger-prick blood test of lipid panel (HDL-cholesterol, triglycerides and LDL-cholesterol) and blood glucose, cognitive function, waist-to-hip ratio, body fat percentages, body mass index respectively and complete a set of psychometric questionnaires, which will take you about 45 minutes, before the interventions (T0), immediately after the 4-week face-to-face intervention (T1) and 12-week after 3-month intervention (T2). The interventions are referring to either MIND, MIND plus FB or usual-care control groups. If you are assigned to MIND group, you will receive four sessions of one-hour nutrition group counselling classes in four consecutive weekdays in a classroom and adoption of MIND for twelve weeks. If you are in MIND plus FB group, you will receive four sessions of two-hour nutrition group counselling classes in four consecutive weekdays in a classroom and four sessions of two-hour forest bathing in four consecutive weekends in a country park. Participants will then be required to self-practice two-hour FB in the country park at daytime at the weekends of 8th week and 12th week of the intervention. If you are in usual-care control, you are required to care as usual. You are also invited to participate a focus group interview after twelve weeks, which will take you about 60 minutes. The focus group interview will be audio-recorded.

# POTENTIAL RISKS/STRESS/PAIN/DISCOMFORTS/OTHER FACTORS AND THEIR MINIMIZATION

The testing should not result in any undue discomfort. The possible minor pain is the finger-prink blood test. Forest bathing will be practiced in a safe place. There will not be encountering any dangerous plants, but we may meet monkeys, bees or insects on this walk. Once you meet them. Stay calm. They will not hurt you. In case of any accident happens, the certified FB guides, who are trained in the wilderness first aid, will provide first aid care to the injured participants.

## POTENTIAL BENEFITS

Participation in this research project is free of charge including nutrition group counselling classes, forest bathing and body measurement tests.

#### PARTICIPATION AND WITHDRAWAL

Document updated date: 20/04/2022

Your participation is voluntary and that you can choose to withdraw from the study at any time you want without any penalty or negative consequences.

#### **CONFIDENTIALITY**

All information related to you will remain confidential and will be identifiable by codes only known to the researchers. The information you provide as part of the project is the research data. Any research data from which you can be identified is known as personal data. Personal data does not include data where the identity has been removed (anonymous data). We will minimize our use of personal data in the study as much as possible. The researcher team will have access to personal data and research data for the purposes of the study. Responsible members of HKMU may be given access to data for monitoring and/or audit of the study to ensure that the research is complying with applicable regulations.

## **QUESTIONS AND CONCERNS**

If you have any questions or concerns about the research study, please feel free to contact Associate Professor, Dr. Queenie Law of HKMU at 3970 2974 or via email: qlaw@hkmu.edu.hk. If you have questions about your rights as a participant of this research study, please contact the Research Ethics Committee of HKMU at 27686251.

## **Consent Form**

Hong Kong Metropolitan University School of Nursing and Health Studies

Effect of Mediterranean-DASH Intervention for Neurodegenerative Delay (MIND) Plus Forest Bathing (FB) on blood pressure and cognitive health for those who are aged 50 and above with hypertension

| I have read and understand the information provided about the above study. I agree to participate in this study. | | |
|---|---|---|
| Name of participant | Signature of participant | Date |
| Name of investigator | Signature of investigator | Date |

Document updated date: 20/04/2022